CLINICAL TRIAL: NCT04143321
Title: Anti-anginal and Antiischemic Effects of Empagliflozin in Diabetic Patients With Refractory Angina:A Phase III, Multicentre, Randomised, Parallel Group, Double Blind Cardiovascular Safety Study of BI 10773 (10 mg Administered Orally Once Daily) Compared to Placebo in Type 2 Diabetes Mellitus Patients With Refractory Angina(EMPT-ANGIN TRIAL)
Brief Title: Antiischemic Effects of Empagliflozin in Diabetic Patients With Refractory Angina
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Masoumeh Sadeghi, professor of cardiology, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EMPT-ANGIN
Record Dates: First submitted 2019-10-13; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus-refractory angina-empagliflozine
MeSH Terms: conditions — Diabetes Mellitus | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- empagliflozin (Experimental): following a two-week washout and complete SAQ and exercise tolerance test patients gave 25 mg empagloflozin and therafter SAQ and ETT was done
  Interventions: Drug: Empagliflozin 25 MG
- No drug (Placebo Comparator): following a two-week washout and complete SAQ and exercise tolerance test patients gave placebo and therafter SAQ and ETT was done
  Interventions: Drug: Empagliflozin 25 MG

INTERVENTIONS:
Drug: Empagliflozin 25 MG — after washout period and EST and SAQ patients gave 25 mg Empagliflozin daily in experimental group

SUMMARY:
this study was aimed to evaluation of antiangial effect of a new fda drug approval on angina in diabetic patient with refractory angina

DETAILED DESCRIPTION:
This was a prospective, double-blind, randomized pilot trial in which a total of 75 subjects were enrolled with T2DM and refractory angina, despite using conventional anti-anginal agents; and were randomly assigned to group A(Empagliflozin group) or B(placebo group) by blinded envelopes method. the study was conducted in two tertiary centers in Isfahan, Iran. The protocol of the study was revised and approved by the institutional ethics committee of Isfahan University of Medical Sciences; and each patient provided an informed consent before participating in the study. The primary aim of the trial was to examine the efficacy of Empagliflozin versus placebo on angina frequency in subjects with T2DM, CAD, and chronic stable angina who remain symptomatic, despite treatment with either one or two anti-anginal agents.The secondary outcome of this study was the evaluation of Physical limitations, angina stability, treatment satisfaction, quality of life, and overall SAQ andeffects o Empaglofolzine vs placebo on treadmill exercise duration, times to angina onset and to 1mm ST segment depression and mean of heart rate recovery(HRR) prior to randomization and after 6 weeks of treatment at peak drug level.

ELIGIBILITY:
Inclusion Criteria:

1- T2DM patients over 18 years of age with CAD, who have had minimum 3-month refractory Angina Pectoris (AP) in spite of using full medical treatment , and were not suitable candidates for revascularization or CABG and reproducible angina, ischemic ST-segment depression of at least 1 mm and limited exercise capacity on treadmill testing (3-9 minutes on a modified Bruce protocol) while receiving full medical treatment .

Exclusion Criteria:

1- New York Heart Association functional class III to IV heart failure symptoms, 2- acute coronary syndrome in the past 2 months, 3-any coronary revascularization during the study period, 4- stroke or transient ischemic attack 5- hepatic or renal impairment, 6-prior treatment with Empagliflozin 7- any relative or absolute contraindication to exercise test or specific condition that preclude accurate interpretation of the electrocardiogram(eg,Left bundle branch block(LBBB),resting ST depression more than 1 mm, pre-excitation or digoxin use).

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Seattle angina questionnaire 1 | 4 weeks
  improvement of angina symptoms

SECONDARY OUTCOMES:
Seattle angina questionnaire 2 | 4 weeks
  evaluation of Physical limitations, angina stability, treatment satisfaction, quality of life, and overall SAQ.
Seattle angina questionnaire 3 | 4 weeks
  evaluation of angina stability,
Seattle angina questionnaire 4 | 4 weeks
  evaluation of treatment satisfaction
Seattle angina questionnaire 5 | 4 weeks
  evaluation of quality of life

OTHER OUTCOMES:
Exercise tolerance test 1 | 4 weeks
  evauation of functional calss Empaglofolzine vs placebo on treadmill exercise duration, times to angina onset and to 1mm ST segment depression and mean of heart rate recovery(HRR)
Exercise tolerance test 2 | 4 weeks
  evaluation of time to angina
Exercise tolerance test 3 | 4 weeks
  evaluation of maximum st depression

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiac rehabilitation research center, Isfahan, Iran